CLINICAL TRIAL: NCT05400759
Title: Clinical Outcomes of the Implementation of Diurnal IOP Curve to 1500 Patients - A Cohort Study.
Status: Completed | Type: Observational
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Diamantis Almaliotis, Dr Sevasti Tsironi, George Papanicolaou Hospital
Other Study IDs: GeorgePH 1500 IOP
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: To Present the Clinical Outcomes of Diurnal IOP Monitoring and Determine Its Value in Our Clinical Practice
Keywords: Tonometric curve, diurnal IOP, IOP phasing, IOP monitoring, glaucoma, glaucoma suspects, IOP peaks, hypertension, compliance, adherence,
MeSH Terms: conditions — Glaucoma; Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IOP monitoring data

SUMMARY:
To present the clinical outcomes of diurnal IOP monitoring and determine its value in our clinical practice.We reviewed the records of 1500 patients (glaucoma suspects or glaucoma patients), who were admitted for diurnal curve during almost 12 years.

DETAILED DESCRIPTION:
We reviewed the records of 1500 patients, who were admitted for diurnal curve during almost 12 years. All patients were hospitalized because their within office-hours exams were considered inadequate and inconclusive for decision-making

744 patients needed change of treatment. 121 patients were programmed for interventional therapy (laser or surgery). 68 patients were declassified, as overdiagnosed and overtreated. In 250 patients hidden adherence problem revealed. In 720 patients peak IOP occurred out of office hours.

ELIGIBILITY:
Inclusion Criteria: IOP diurnal curve consisted of glaucoma patients with intraocular pressure higher than target pressure despite referred previously sufficient therapy and also patients with equal or lower than target pressure, but with disease progression. There were also included patients with advanced glaucoma with visual field defects on the visual field testing, as well as patients with normal tension glaucoma and labile secondary glaucomas (exfoliative, pigmentary and chronic angle closure glaucoma), for whom close monitoring and therapy reconsidering was judged appropriate.Glaucoma suspects, demonstrating findings consistent with increased risk for glaucoma development, were included.

-

Exclusion Criteria: Patients with missing data values for IOP

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were retrieved from the eye clinic database. The records of all 1500 patients were retrospectively reviewed. We included the last 1500 patients who had undergone diurnal IOP monitoring in the clinic until the conduct of the study. All of them were hospitalized between November 2007 and December 2019, at the Eye Clinic of General Hospital "George Papanikolaou" in Thessaloniki, Greece.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Diurnal IOP monitoring | 12 years
  This analysis provides a "real life' account of IOP in a large number of glaucoma suspects and patients. Our results demonstrate the potential for significant additional information, being obtained from diurnal IOP monitoring, in clinical practice.

IPD SHARING:
Plan to Share IPD: No